CLINICAL TRIAL: NCT05628545
Title: Clinical Study on Adoptive Treatment of Advanced Hepatocellular Carcinoma With Allogeneic γδ-T Cells
Brief Title: Adoptive Treatment of Advanced Hepatocellular Carcinoma With Allogeneic γδ-T Cells
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: COVID1-19 pandemic
Sponsor: Guangdong GD Kongming Biotech LLC (Industry)
Collaborators: Jinan University Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GDKM-100-08HEP
Record Dates: First submitted 2022-11-02; First posted 2022-11-28 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; gamma delta T cell; Allogeneic; Adoptive Treatment
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GDKM-100 injection (Experimental): In this trial, the patients will receive multiple high-activity γδ T cell immunotherapies.The trial is divided into two parts: Part 1 is a multiple-dose escalation trial consisting of 3 dose groups (2×10^8 cells/person, 5×10^8 cells/person, 10×10^8 cells/person at 1-3 infusion, 4-6 infusion and 7-9 infusion), with 9 patients planned to be enrolled. Part 2 is a single dose trial in which doctor and the PI evaluates whether to give the rest patients to receive the 10×10^8 cells/person infusions based on available safety data.
  The check indexes are CT scan，intestinal flora detection and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Biological: GDKM-100 injection

INTERVENTIONS:
Biological: GDKM-100 injection — Participants will received GDKM-100injection (allo-γδ T Cells) Infusion every two weeks.

SUMMARY:
Brief Summary: In this study, effects of γδ T cells on Advanced hepatocyte carcinoma The goal of this clinical trial is to learn about effects of allogeneic γδ T therapy in advanced hepatocyte carcinoma patients.

The main question it aims to answer is:Will advanced hepatocyte carcinoma patients be benefit from allogeneic γδ T therapy? Participants will received GDKM-100injection (allo-γδ T Cells) Infusion every two weeks.

ELIGIBILITY:
Inclusion criteria

1. Age is 18-75 years old, and gender is unlimited;
2. HCC was confirmed by pathological or clinical examination;
3. Patients with stage CNLCIII, IV primary HCC who are receiving second-line treatment / unable to receive existing treatments, or CNLCI and II of primary HCC patients who are unable to receive existing treatments;
4. Male subjects with partner women of childbearing age must have reliable, effective methods of contraception starting from the signing of the informed consent form until 120 days after the last dose of the study drug. Male subjects with a pregnant spouse must use condoms without other contraceptive methods;
5. Participants volunteered to join the study, signed an informed consent, had good compliance, and cooperated with the follow-up.

Exclusion criteria

1. Gastrointestinal bleeding, refractory ascites, hepatic encephalopathy, or hepatorenal syndrome;
2. Accept other cellular or immune clinical experiments within 8 weeks before enrollment;
3. Immunological deficiency, a known immunosuppressive disease or HIV;
4. Active infection, unexplained fever;
5. Serious or unstable heart, lung, kidney and hematopoietic system diseases;
6. Autoimmune diseases, such as rheumatoid arthritis;
7. Neurological diseases, diffuse leptomeningeal diseases; combined with neurodegenerative diseases;
8. Hormone use during cell therapy: dexamethasone dose exceeds 2mg / day during immunotherapy;
9. Pregnant or lactating women;
10. The subject had a known history of psychotropic substance abuse or drug use; he had stopped drinking Patients can be enrolled; 11 In the judgment of the investigator, the subject has other factors that may cause the forced termination of the study, such as other serious diseases or serious abnormal laboratory examination or other family or social factors that will affect the subject's safety of the subject, or the collection of trial data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
The change of performance status score | up to approximately 16months
  In medicine(oncology and Other fields), performance status is an attempt to Quantify cancer patients' general well-being and activities of daily life.This measure is used to determine whether they can receive chemotherapy, whether dose adjustment is necessary，and as a measure for the required intensity of palliative care. It is also used in oncological randomized controlled trials as a measure of quality of life.
  PS scores range from 1 to 5,with Higher PS score indicating worse prognosis.
The Child-Pugh score | up to approximately 16months
  The Child-Pugh score is a system for assessing the prognosis-including the required strength of treatment and necessity of liver transplant-of chronic liver disease. It provides a forecast of the increasing severity of liver disease and expected survival rate.Child-Pugh scores range from 5 to 15, with higher scores indicating worse prognosis.Class A: 5-6, Class B: 7-9, Class C: 10-15 (minimum 5, maximum 15;)
Overall Survival | Up to 16months
  From the date of entry into the clinical study until death from any cause

SECONDARY OUTCOMES:
ORR（objective remission rate ） | up to approximately 16months
  ORR is defined as the percentage of participants in the analysis population who have a Complete Responseor a Partial Response .
  CR: Disappearance of all target lesions PR: at least 30% decrease in the sum of diameters of target lesions
TTP（time to disease progression ) | up to approximately 16months
  Time to progression is defined as the time from study enrollment until radiological progression in a previously embolized lobe, development of new lesions in an untreated lobe, or evidence of extrahepatic progression .Patients that die of causes unrelated to the study drug without evidence of progression will be censored. Participants without progression at the time of analysis were censored at their last date of tumor evaluation.
DoR(duration of remission ) | up to approximately 16months
  The duration of response (DoR) is measured from the time the criteria are met for CR or PR (whichever is first recorded) until the date that recurrent or progressive disease is documented.
  CR: Disappearance of all target lesions PR: at least 30% decrease in the sum of diameters of target lesions
DCR (disease control rate) | up to approximately 16months
  DCR is defined as the percentage of participants in the analysis population who have a CR, PR or SD.
  CR(complete response)：Disappearance of all target lesions PR( partial response)：at least 30% decrease in the sum of diameters of target lesions SD(stable disease）：any cases that do not qualify for either partial response or progressive disease.
PFS（Progression-Free Survival ) | up to approximately 16months
  Progression-Free Survival (PFS) is defined as the duration of time from start of treatment to time of objective disease progression or death from any cause without evidence of disease progression, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi nan Yin, PhD.MD., Principal Investigator — Jinan University
Locations (1):
- Zhuhai People'S Hospital, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No